CLINICAL TRIAL: NCT01399515
Title: Efficacy and Safety of Oral Valproic Acid for Retinitis Pigmentosa
Acronym: VPA_RP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong Gon Yu, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH_OT_VPA
Record Dates: First submitted 2011-05-03; First posted 2011-07-21 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Eye Disease, Hereditary; Retinal Degeneration
Keywords: Retinitis pigmentosa; Valproic acid
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Degeneration | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valproic acid (Active Comparator)
  Interventions: Drug: Valproic Acid
- Control (No Intervention)

INTERVENTIONS:
Drug: Valproic Acid — One 500mg tablet by mouth daily
  Other Names: Valproate
  Arms: Valproic acid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of oral valproic acid to slow the progression of visual function and/or to improve the visual function in patients with retinitis pigmentosa (RP).

Enrolled subjects in valproic acid group will be treated with oral valproic acid 500mg daily for 48 weeks. Visual function and safety will be assess before and after treatment (48 weeks) between valproic acid and control groups.

DETAILED DESCRIPTION:
This study is designed as a single-site, interventional, prospective, non-randomized, controlled study of 200 participants. Patients that participate in the study will be assigned to either valproic acid group or control in a 3:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of retinitis pigmentosa (RP) established by night blindness, visual field constriction, marked reduction of electroretinogram, and the clinical signs of RP in fundus examination
* Best corrected visual acuity of 20/200 or more on a Snellen chart in at least one eye
* Intact visual field of 5 or more as measured by the kinetic perimetry
* Understand and sign the IRB-approved informed consent document for the study
* Body weight: male (40 kg to 100 kg), female (40 kg to 80 kg)
* Must be able to swallow tablets
* Female subjects of childbearing potential must commit to practice acceptable methods of contraception

Exclusion Criteria:

* Pregnant women
* Lactating mothers
* Medical problems that make consistent follow-up over the treatment period unlikely (e.g., stroke, myocardiac infarction, malignancy) or severe systemic disease
* Other ocular disease: retinal disease other than RP or cystoid macular edema, glaucoma, cataract worse than +2PSC or infectious corneal disease
* Coagulation disorder or bleeding-tendency
* Liver dysfunction
* Renal dysfunction
* History of pancreatitis
* History of neurological disorders including epilepsy, history of brain injury or any organic brain disorders
* History of mental disorders including schizophrenia, bipolar disorder, or suicidality
* Currently receiving valproic acid or other anti-convulsants
* Has taken one of the following drugs at least 4 weeks prior to enrollment as these drugs are specifically known to affect the progression of RP: vitamin A, lutein, omega-3 fatty acid, or any antioxidant which affect the blood flow of retina or retinal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mean change in visual field area from baseline to 48 weeks | Baseline, week 24, and week 48
  Visual field area will be measured using kinetic perimetry (Goldmann perimetry) or static perimetry including the central 30 field.

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) | Baseline, week 24, and week 48
  BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS)
Mean change in 30-Hz flicker Electroretinogram (ERG) amplitude | Baseline and week 48
Mean change in central macular thickness | Baseline, week 24, and week 48
  Central macular thickness as measured by Optical Coherence Tomography (OCT)
Mean change in fundus appearance | Baseline and week 48
  Fundus appearance as judged by color fundus photography
Mean change in total score on vision-related quality of life | Baseline and week 48
  Total score on vision-related quality of life as measured by the National Eye Institute Visual Function Questionnaire (NEI-VFQ25)
Occurrence of adverse effect related to Valproic acid | Baseline through 48 weeks
Changes in clinical laboratory data | Baseline through 48 weeks
  CBC, BUN, Creatinine, Liver panel (Cholesterol, Total protein, Albumin, Total bilirubin, Alkaline phosphatase, AST, ALT, GGT), Coagulation panel (PT INR, PT%, PT sec, aPTT, Fibrinogen), Electrolyte panel (Na, K, Cl, TCO2)
Mean change in central macular volume | Baseline, week 24, and week 48
  Central macular volume as measured by Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Gon Yu, MD, PhD, Principal Investigator — Department of Ophthalmology, Seoul National University Hospital
Locations (1):
- Department of Ophthalmology, Seoul National University Hospital, Seoul, South Korea